CLINICAL TRIAL: NCT01287715
Title: When and in Whom to Stop Etanercept After Successful Treatment of Juvenile Idiopathic Arthritis
Brief Title: Withdrawal of Etanercept After Successful Treatment of Juvenile Idiopathic Arthritis
Acronym: ABC-STOP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Dutch Arthritis Association (Industry)
Responsible Party: L.W.A. van Suijlekom-Smit, MD, PhD, MSCE, Erasmus Medical Center Sophia Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NR 10-1-203
Record Dates: First submitted 2011-01-31; First posted 2011-02-01 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2011-01

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- STOP-arm (Experimental): Discontinuation of etanercept
  Interventions: Drug: etanercept
- CONTROL-arm (No Intervention): Continuation of etanercept for another 9 months, and, if still meeting the eligibility criteria, discontinuation of etanercept thereafter.
  Interventions: Drug: etanercept

INTERVENTIONS:
Drug: etanercept — Discontinuation of etanercept (half of the dosis for 3 months and discontinuation thereafter)
  Other Names: enbrel
  Arms: STOP-arm
Drug: etanercept — Continuation of etanercept for another 9 months, and, if still meeting the eligibility criteria, discontinuation of etanercept thereafter.
  Other Names: enbrel
  Arms: CONTROL-arm

SUMMARY:
The purpose of this study is to determine whether etanercept can be withdrawn successfully (i.e. no occurrence of flares) in juvenile idiopathic arthritis (JIA) patients in whom disease remission is reached.

Goals:

1. to investigate in a randomized controlled trial:

   * which proportion of JIA patients in remission can successfully discontinue etanercept compared to JIA patients in remission who continue etanercept;
   * if time in remission on etanercept is an important factor in retaining remission after discontinuation of etanercept.
2. to investigate in alle JIA patients who discontinue etanercept (including the control group):

   * predicting factors (patient or disease characteristics, including time in remission, and MRP8/MRP14) for successfully discontinuation of etanercept;
   * the disease course after discontinuation of etanercept (time to flare) and the effect of restarting etanercept after flaring.

DETAILED DESCRIPTION:
Juvenile Idiopathic Arthritis (JIA) is the most common cause of chronic arthritis in children. Etanercept has proven to be an effective treatment for JIA. Considering the risk of occurrence of long-term side-effects and to prevent the burden of the weekly injections and costs, it is a logical step to discontinue etanercept after reaching remission (no disease activity for at least six months). Especially since there are concerns about the long-term effect of suppressing the immune system with etanercept. However, little is known about if successful discontinuation is possible or when to stop. Risk is that the disease might flare (reactivate) again.

For this study, JIA patients in remission will be selected from the ABC-register (an observational study including all Dutch JIA patients who use etanercept). Eligible patients will be randomized to stop etanercept or continue it for another 9 months. Patients are followed with standard visits evaluating disease activity until 12 months after discontinuation of etanercept. In case of a disease flare etanercept therapy will be reintroduced immediately and the patient will be treated according to the insight of their treating physician. Expected is that JIA patients who were in remission for more than 12 months before discontinuation have a better chance to retain remission.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Juvenile Idiopathic Arthritis (all subtypes) by the International League of Associations of Rheumatology (ILAR) criteria
* On etanercept therapy
* No MTX or low dose MTX (maximum 10 mg/m2)
* 3 or more months in remission according to the criteria of Wallace (i.e. 9 or more months of inactive disease)
* Age ≥4 and <18 years at start of study
* Written informed consent from parents and patients 12 years and over

Exclusion Criteria:

* Systemic corticosteroids (up to 9 months prior to inclusion)
* Intra-articular corticosteroids (up to 6 months prior to inclusion)
* Synthetic DMARDs besides low dose MTX (up to 9 months prior to inclusion)
* Biologic DMARDs besides etanercept (up to 9 months prior to inclusion)

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Flare-rate | 9 months
  To evaluate if the flare-rate is different between the 2 arms (continuation and discontinuation of etanercept).

SECONDARY OUTCOMES:
Duration of remission before withdrawal of etanercept | 9 months
  To evaluate between the 2 arms (continuation and discontinuation of etanercept) if time in remission on etanercept is an important factor in retaining remission after discontinuation of etanercept.
Predictors for successful discontinuation of etanercept | 12 months after discontinuation of etanercept
  Evaluation of predictors (patient or disease characteristics, including time in remission, and MRP8/MRP14) for successful discontinuation of etanercept in all JIA patient who discontinue etanercept.
Disease course after flaring | 6 months after flare
  After a flare (exacerbation) occurs: evaluation of time to flare and the effect of restarting etanercept after flaring.

CONTACTS AND LOCATIONS:
Overall Officials: LWA van Suijlekom-Smit, MD,PhD,MSCE, Principal Investigator — Erasmus Medical Center
Locations (10):
- Netherlands (10):
  - Academic Medical Centre Emma Children's Hospital, Amsterdam
  - Reade Institute Amsterdam, Amsterdam
  - Sint-Lucas Andreas Hospital, Amsterdam
  - University Medical Centre Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Maastricht University Medical Centre, Maastricht
  - St Maartenskliniek, Nijmegen
  - Erasmus MC Sophia Children's Hospital, Rotterdam
  - Haga Hospital, Juliana Children's Hospital, The Hague
  - Utrecht Medical Centre Wilhelmina Children's Hospital, Utrecht